CLINICAL TRIAL: NCT04321993
Title: Treatment of Moderate to Severe Coronavirus Disease (COVID-19) in Hospitalized Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lisa Barrett (Other)
Collaborators: Nova Scotia Health Authority (Other); Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Lisa Barrett, Clinician Scientist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAIL-004
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: COVID; coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — baricitinib; Janus Kinase Inhibitors; remdesivir; Antiviral Agents; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Baricitinib (Experimental): Moderate and severe, not critical disease
  Interventions: Drug: Baricitinib (janus kinase inhibitor)
- Remdesivir (Experimental): Moderate and severe, not critical disease
  Interventions: Drug: Remdesivir (antiviral)
- Remdesivir + baricitinib (Experimental): Moderate and severe, not critical disease
  Interventions: Drug: Remdesivir (antiviral) + barictinib (janus kinase inhibitor)
- Tocilizumab (Experimental): Severe, critical disease
  Interventions: Drug: Tocilizumab (interleukin 6 inhibitor)
- Clinical standard of care (No Intervention): Moderate and severe, not critical disease AND severe, critical disease as applicable

INTERVENTIONS:
Drug: Baricitinib (janus kinase inhibitor) — Baricitinib will be administered as 4 mg po daily for 14 days or until hospital discharge, whichever is sooner.
  Arms: Baricitinib
Drug: Remdesivir (antiviral) + barictinib (janus kinase inhibitor) — Remdesivir will be administered as a loading dose of 200 mg IV over one hour on day 1 followed by 100 mg IV daily over one hour on days 2-5 (with a possibility to extend to up to 10 days total).
  Baricitinib will be administered as 4 mg po daily for 14 days or until hospital discharge, whichever is sooner.
  Arms: Remdesivir + baricitinib
Drug: Remdesivir (antiviral) — Remdesivir will be administered as a loading dose of 200 mg IV over one hour on day 1 followed by 100 mg IV daily over one hour on days 2-5 (with a possibility to extend to up to 10 days total).
  Arms: Remdesivir
Drug: Tocilizumab (interleukin 6 inhibitor) — Tocilizumab will be administered as a single IV infusion over one hour. Dosage will be 8 mg/kg total bodyweight up to a maximum of 800 mg.
  Arms: Tocilizumab

SUMMARY:
Investigational medications adjunct to clinical standard of care treatment will be assessed to evaluate safety and effectiveness as an anti-COVID-19 treatment. All hospitalized persons with moderate to severe COVID-19 disease that meet eligibility criteria will be offered participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Moderate to severe COVID-19 associated disease as defined by the WHO
* Willing and able to provide informed consent prior to performing study procedures
* Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay
* Illness of any duration, and at least one of the following: Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), or Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤ 94% on room air, or Require mechanical ventilation and/or supplemental oxygen.
* Normal potassium, magnesium, and calcium levels pre-therapy when used in agents at risk of QT prolongation

Patients will be further distinguished based on their disease severity into one of two categories:

* Moderate and severe, not critical disease: patients with SpO2 ≤ 94% on room air, and those who require supplemental oxygen
* Severe, critical disease: patients with critical illness requiring ICU-level care including requiring mechanical ventilation or ECMO, and/or end organ dysfunction as seen in sepsis/septic shock.

Exclusion Criteria:

* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN)
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive study treatment Medication specific Exclusion

Baricitinib:

1. Contraindicated for patients with known hypersensitivity to baricitinib or to any of the excipients.
2. Prior untreated latent tuberculosis
3. Any individuals with TB risk factors will not be enrolled in the baricitinib arm of the study.
4. Presence of active viral hepatitis C or B
5. People with a clinical history of invasive or active fungal infection
6. People with a clinical history of active CMV disease in the last year
7. Patients who are pregnant or breastfeeding
8. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR <15)

Tocilizumab:

1. Known hypersensitivity to tocilizumab or any of its components
2. Prior untreated latent tuberculosis
3. Any individuals with TB risk factors will not be enrolled in the tocilizumab arm of the study.
4. Presence of active viral hepatitis C or B
5. People with a clinical history of invasive or active fungal infection
6. People with a clinical history of active CMV disease in the last year
7. CRP<75 mg/L
8. SpO2 ≥ 92% on room air

Remdesivir:

1. Known hypersensitivity to remdesivir or any of its components
2. Weight below 40 kg
3. SpO2 ≥ 94% on room air
4. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. eGFR <30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Clinical status of subject at day 15 (on a 7 point ordinal scale). | Up to 15 days
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.

SECONDARY OUTCOMES:
Status on an ordinal scale assessed daily while hospitalized and on days 15 and 29 and 180. | Up to 180 days
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or ECMO;
  7. Death.
Length of time to clinical improvement | Up to 29 days
  Time to clinical improvement is defined as the time to normalization of respiratory rate, fever, and oxygen saturation, and alleviation of cough within 72 hours.
Number of participants with normal pulmonary function and normal O2 saturation on days 11, 15 and 29 | Up to 29 days
Number of participants that developed Acute Respiratory Distress Syndrome (ARDS) after treatment | Up to 24 weeks
Length of time to clinical progression | Up to 29 days
  Time to clinical progression, defined as the time to death, mechanical ventilation, or ICU admission
Cause of death (if applicable) | Up to 24 weeks
Sequential Organ Failure Assessment (SOFA) score, daily while hospitalized and on days 15 and 29. (Initial, highest, deltas and mean) | Up to 29 days
Length of time to normalization of fever | Up to 29 days
  Fever normalization as defined by: Temperature < 36.6 °C armpit, < 37.2 °C oral, or < 37.8 °C rectal sustained for minimum 24 hours
Length of time to normalization of oxygen saturation | Up to 29 days
  Oxygen normalization as defined by: peripheral capillary oxygen saturation (Sp02) > 94% sustained minimum 24 hours.
Duration of supplemental oxygen (if applicable) | Up to 29 days
Duration of mechanical ventilation (if applicable) | Up to 29 days
Duration of hospitalization | Up to 29 days
Adverse events | Up to 180 days

OTHER OUTCOMES:
Global and SARS-CoV-2-specific immune responses before, during and after intervention and in standard of care treatment arm | Up to 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada